CLINICAL TRIAL: NCT01495442
Title: Evaluation of a Dry Powder Aerosol Dispersion Mechanism by Radiolabeling Techniques
Acronym: DPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, William Bennett, PhD, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 11-1260
Record Dates: First submitted 2011-12-12; First posted 2011-12-20 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Adult Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified Handihaler DPI (Active Comparator)
  Interventions: Device: modified Handihaler DPI
- standard Handihaler DPI (Placebo Comparator)
  Interventions: Device: standard Handihaler DPI

INTERVENTIONS:
Device: modified Handihaler DPI — subjects randomized to receive 1 inhaled dose on 2 separate days, each dose delivered 2-3 days apart. The radiolabeled albuterol drug powder will be dispersed from either the DET bead-HandiHaler prototype or via the established HandiHaler device standard with the lactose-albuterol formulation provided to us by the sponsor.
  Arms: modified Handihaler DPI
Device: standard Handihaler DPI — subjects randomized to receive 1 inhaled dose on 2 separate days, each dose delivered 2-3 days apart. The radiolabeled albuterol drug powder will be dispersed from either the DET bead-HandiHaler prototype or via the established HandiHaler device standard with the lactose-albuterol formulation provided to us by the sponsor.
  Arms: standard Handihaler DPI

SUMMARY:
The primary objective is to admix a radiolabel with albuterol sulphate for incorporation into the Handihaler® device for inhalation studies. This will allow for the investigators to determine the regional lung deposition of drug inhaled from the standard Handihaler® device compared to a novel modification of the device to provide more effective dispersion and aerosolization of the coated albuterol powder. The new mechanism of action for proof-of-concept testing consists of a bead (5.1 mm; expanded polystyrene foam) coated with drug powder, as opposed to the standard lactose formulation-filled capsule.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers adults

Exclusion Criteria:

* chronic illness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Fractional delivery of dry powder to the lung | 1-5 minutes post inhalation
  To compare the in vivo performance,i.e. the fraction of drug loaded in device that is delivered to the lung, of the novel system in comparison with a standard marketed dry powder inhaler (DPI) using radio-imaging techniques. The fraction delivered to the lung will be determined by gamma camera imaging of the lungs following inhalation of the radiolabeled powder from the standard vs. new device.

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, CEMALB, Chapel Hill, North Carolina, United States